CLINICAL TRIAL: NCT05215184
Title: Defense Health Agency- Development of a Medical Device Utilizing an EEG-Based Algorithm for the Objective Quantification of Pain
Acronym: PQXDOD1
Status: Completed | Type: Observational
Sponsor: PainQx, Inc (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: Pro00054666
Record Dates: First submitted 2022-01-17; First posted 2022-01-31 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Chronic Pain Patients
  Interventions: Device: Zeto WR19 EEG Recording
- Healthy Controls
  Interventions: Device: Zeto WR19 EEG Recording

INTERVENTIONS:
Device: Zeto WR19 EEG Recording — 15 minutes of EEG recording to be obtained from eligible participants

SUMMARY:
PainQx, with the support of the Department of Defense (Contract #W81XWH-21-C-0034), is conducting a study to collect electroencephalography (EEG) data from people with chronic pain in order to develop algorithms than will objectively assess the pain a person is experiencing. EEG is a monitoring method that records electrical activity in the brain. If enrolled in the study, subjects will be asked to answer a series of questions regarding their level of chronic pain, level of functionality, symptoms, behavioral health information, and medications, and subsequently have a 15 minute, non-invasive EEG recording taken by placing electrodes along the scalp. Through participation, chronic pain subjects will provide data needed to further develop this technology.

ELIGIBILITY:
Inclusion Criteria:

* Male and female chronic pain patients
* Patients between the ages of 18-85 years
* Patients exhibiting the presence of symptoms in excess of 3 months duration
* Patients suffering from neuropathic (e.g., lower back pain), osteoarthritis, or muscular skeletal pain
* Patients with evidence of pathology related to the painful condition on which diagnosis was made (e.g., results of imaging or diagnostic pain code)
* Patients with NRS pain scores across the full range (0-10) at the time of testing

Exclusion Criteria:

* • Patients with medically diagnosed psychotic illness, such as Schizophrenia

  * Patients with medically diagnosed drug or alcohol dependence in the past 12 months
  * Patients with a medical history of head injury with loss of consciousness and amnesia (within the last 2 years)
  * Patients with skull abnormalities that preclude the proper placement of the electrodes for EEG data acquisition
  * Patients who have a spinal cord stimulator, neurological implants, deep brain stimulators, or other pain related implantable devices such as an intrathecal drug pump
  * Patients for whom the source of pain at the time of the evaluation is associated with: neurological disorders (multiple sclerosis, Parkinson, dementia), diabetes, migraines, or those with reflex / sympathetic dystrophy disorder/complex regional pain syndrome, fibromyalgia, or visceral pain

    o Note: This does not exclude patients who suffer from these disorders if the current source of pain is not due to the disorder. For example, patients with diabetes are NOT excluded, but patients whose pain at the time of the evaluation is a result of diabetic neuropathy are excluded. Similarly, patients with a history of migraines but for whom a migraine is not the current source of pain at the time of the evaluation are NOT excluded.
  * Patients with cancer

    o Note: This does not exclude patients who have been in complete remission for more than two years
  * Patients on workers compensation or disability or have other circumstances which may cause/incentive them to misreport their pain
  * Patient on gabapentin or pregabalin (within the last month)
  * Patients on experimental drugs (i.e. participating in drug trial), use off-label drugs, or are on unapproved dosages
  * Patients who have a history of seizures (within the past 3 months)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A minimum of two hundred twenty-five (225) male and female chronic pain patients between the ages of 18-85 years will be enrolled in the study. A minimum of seventy-five (75) healthy normal subjects between the ages of 18-85 years will also be enrolled. The normal subjects are added to assure that the study spans the entire pain scale including those with a self-reported pain score of 0. Subjects who meet inclusion/exclusion criteria will be asked to participate and to provide informed consent. The study will enroll up to 350 patients.
Sampling Method: Non-Probability Sample
Enrollment: 278 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Pearsons Correlation between ALGOS derived pain biomarker and patient reported Defense and Veterans Pain Rating Scale (0-10) | Data analysis occurs within 3 months of study completion

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Panorama Orthopedics & Spine Center, Golden, Colorado
  - Indiana Spine Group, Carmel, Indiana
  - Comprehensive Spine and Pain Center of New York, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Center for Interventional Pain and Spine, Lancaster, Pennsylvania

IPD SHARING:
Plan to Share IPD: No